CLINICAL TRIAL: NCT03891927
Title: Effect of Extra Virgin Olive Oil on Glycemic Control ,Insulin Resistance and Insulin Secretion in Patients With Type 2 Diabetes
Brief Title: Extra Virgin Olive Oil on Glycemic Control ,Insulin Resistance and Insulin Secretion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aml Ali Aboelghait, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: olive oil on glycemic control
Record Dates: First submitted 2019-03-18; First posted 2019-03-27 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Insulin Resistance
Keywords: olive oil; glycemic control
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Intervention Model Description: randomized clinicl trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- olive group (Experimental): During the experimental period (3 months ), participants will be requested to consume daily dose of 30 mL (3 tablespoons) of HP-EVOO ( high polypheol Extra virgin olive oil)
  Interventions: Dietary Supplement: extra virgin olive oil
- non olive group (No Intervention): No intervention

INTERVENTIONS:
Dietary Supplement: extra virgin olive oil — During the experimental period (3 months ), participants will be requested to consume daily dose of 30 mL (3 tablespoons) of HP-EVOO
  Arms: olive group

SUMMARY:
Aim of this study to evaluate the effects of extra virgin olive oil on glycemic control ,insulin resistance and insulin secretion in patients with Type 2 diabetics.

DETAILED DESCRIPTION:
Diabetes is a major health problem and one of the leading causes of morbidity and mortality worldwide. Lifestyle and particularly dietary habits are considered key issues in both the prevention and management of the disease aimed at achieving an adequate glycemic control or at delaying the onset of diabetic chronic complications .

Olive oil (OO) has been recognized for centuries for its nutritional properties and considered as the "elixir of youth and health" by antique Greeks. Extra virgin olive oil is the main source of dietary fat in the Mediterranean diet . Consumption of extra virgin olive oil might exert beneficial effects in the prevention, development and progression of T2D compared with refined olive oil .

Several bioactive ingredients within OO have been repeatedly linked with anti-oxidant and anti-inflammatory preventative functions, particularly those from monounsaturated fatty acids (MUFA), and key biophenols such as oleuropein and hydroxytyrosol (HT) . Biophenols may influence glucose metabolism via several mechanisms; inhibition of carbohydrate digestion and glucose absorption in the intestine, activation of insulin receptors and glucose uptake in the tissues, antioxidative properties, potent free-radical scavenging and immunomodulatory effects. Multiple studies proven that EVOO improve metabolic control by affection of adipokines .The inhibition of carbohydrate digestion and absorption takes place through an inhibition of some digestive enzymes, especially the carbohydrate-hydrolyzing enzymes α-amylase and α glucosidase. Inhibition of these enzymes retards carbohydrate digestion, thus causing a reduction in glucose absorption rate .With their antioxidative properties, polyphenols diminish the production of advanced glycosylated end products such as HbA1c, AGEs, which are readily formed and accumulated with sustained hyperglycemia, contribute to the development of diabetic complications. As a consequence, inhibition of AGE formation constitutes an attractive therapeutic/preventive target .

Studies both in healthy subjects and in persons with type 2 diabetes mellitus have demonstrated that levels of GLP-1are increased more by dietary MUFA than by dietary saturated fatty acids, and that the greater postprandial clearance of an oral overload of MUFA-rich fats is associated with a greater increase in postprandial incretins such as GLP-1 or gastric inhibitory polypeptide. MUFAs from olive oil, therefore, appear to significantly increase the insulin and GPL-1 secretion .

ELIGIBILITY:
Inclusion Criteria:

- Patients with type 2 diabetes with

* age 30-60 years regardless of their gender.
* Duration of diabetes less than 5 years.
* on oral antihyperglycemic medication.
* willing to participate in research.

Exclusion Criteria:

* Type 1 diabetes.
* Insulin treated type 2 DM patients.
* Pregnant women .
* Patients on cholesterol-lowering drugs, steroids and other drugs that affect the fat metabolism.
* Patients on regular (days) supplement that contain olive oil.
* Patients have aversion or allergy to olive oil.
* Smokers .
* Patients have gall bladder disease ,gastrointestinal disease (e.g.malabsorption),liver,kidney,heart and thyroid diseases.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
change of HBa1c (glycated hemoglobin) after intervention by extra virgin olive oil | 3 months
  change of HBa1c (glycated hemoglobin) after intervention by 30 ml extra virgin olive oil daily for three months and comparison that with other group (no intervention of olive oil) to evaluate glycemic control .
  measurment of HBa1c for group of intervention at baseline and after 3 months intervention .
  and other group (no intervention of olive oil) at baseline and after 3 months.
change of fasting glucose after intervention by extra virgin olive oil | 3 months
  change of fasting glucose after intervention by 30 ml extra virgin olive oil daily for three months and comparison that with other group (no intervention of olive oil) to evaluate glycemic control .
  measurment of fasting glucose for group of intervention at baseline and after 3 months intervention .
  and other group (no intervention of olive oil) at baseline and after 3 months.

SECONDARY OUTCOMES:
calculating of insulin resistance and insulin secretion after intervention by extra virgin olive oil | 3 months.
  measurement of fasting insulin after intervention by 30 ml extra virgin olive oil daily for three months and comparison that with other group (no intervention of olive oil) to evaluate insulin resistance and insulin secretion by calculating HOMA -IR and HOMA-B The HOMA-beta cell function (HOMA-B) will be calculated by using the following formula: 360 x fasting insulin (μU/mL) / (fasting glucose (mg/dL) - 63).
  (HOMA-IR) method: fasting glucose (mg/dl) x fasting insulin / 405
reduction of systolic and diastolic blood pressure after intervention by extra virgin olive oil . | 3 months
  measurement of systolic and diastolic blood pressure after intervention by 30 ml extra virgin olive oil daily for three months and comparison that with other group
reduction of body mass index . | 3 months
  height , weight measuring and calculating BMI.Body mass index (BMI) was calculated as weight (kg) divided by squared height (m).
changing in waist circumference . | 3 months follow up
  waist circumference change will be measured by tape measure at the umbilical level while patients standing after expiration by centimeter after intervention by 30 ml extra virgin olive oil daily for three months
change at Lipid profile (cholesterol, TG, LDL, HDL) after intervention . | 3 months follow up
  change at Lipid profile (cholesterol, TG, LDL, HDL) (cholesterol by mg/dl ,triglyceride by mg/dl ,low density lipoprotein by mg/dl and high density lipoprotein by mg/dl ) after intervention by 30 ml extra virgin olive oil daily for three months and comparison that with other group (no intervention of olive oil)

CONTACTS AND LOCATIONS:
Overall Officials: Salah Abdelazeem Argoon, professor, Study Director — Assiut University

REFERENCES:
- [Background] Schwingshackl L, Lampousi AM, Portillo MP, Romaguera D, Hoffmann G, Boeing H. Olive oil in the prevention and management of type 2 diabetes mellitus: a systematic review and meta-analysis of cohort studies and intervention trials. Nutr Diabetes. 2017 Apr 10;7(4):e262. doi: 10.1038/nutd.2017.12. PMID 28394365
- [Background] Santangelo C, Filesi C, Vari R, Scazzocchio B, Filardi T, Fogliano V, D'Archivio M, Giovannini C, Lenzi A, Morano S, Masella R. Consumption of extra-virgin olive oil rich in phenolic compounds improves metabolic control in patients with type 2 diabetes mellitus: a possible involvement of reduced levels of circulating visfatin. J Endocrinol Invest. 2016 Nov;39(11):1295-1301. doi: 10.1007/s40618-016-0506-9. Epub 2016 Jun 25. PMID 27344308
- [Background] Nigam P, Bhatt S, Misra A, Chadha DS, Vaidya M, Dasgupta J, Pasha QM. Effect of a 6-month intervention with cooking oils containing a high concentration of monounsaturated fatty acids (olive and canola oils) compared with control oil in male Asian Indians with nonalcoholic fatty liver disease. Diabetes Technol Ther. 2014 Apr;16(4):255-61. doi: 10.1089/dia.2013.0178. PMID 24625239
- [Background] Lama A, Pirozzi C, Mollica MP, Trinchese G, Di Guida F, Cavaliere G, Calignano A, Mattace Raso G, Berni Canani R, Meli R. Polyphenol-rich virgin olive oil reduces insulin resistance and liver inflammation and improves mitochondrial dysfunction in high-fat diet fed rats. Mol Nutr Food Res. 2017 Mar;61(3). doi: 10.1002/mnfr.201600418. Epub 2016 Dec 20. PMID 27794174